CLINICAL TRIAL: NCT05816811
Title: Power Exercise for Stroke Recovery: The POWER Feasibility Trial
Acronym: POWER-F
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Ada Tang, Associate Professor, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POWER Feasibility
Record Dates: First submitted 2023-03-20; First posted 2023-04-18 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Stroke
Keywords: Stroke; Resistance training; Power training; Feasibility study; Skeletal muscle
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Single-group pilot trial aimed at examining the feasibility of a 10-week power-focused resistance training intervention for people with stroke
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Power Training (Experimental): The program is intentionally designed with 3 progressive phases: Phase 1 Familiarization (Week 1) will allow participants to begin with a low-intensity version of the training program (body weight resisted or light weights at RPE 2-3 for 8 repetitions) to acclimate participants to the movements. Phase 2 Strength (Weeks 2-5) will progress in loads to achieve volitional fatigue between 5-8 repetitions (RPE 7-9). Phase 3 Power (Weeks 6-10) will use intensities between RPE 4-6 (15-20 repetitions) and execute each exercise at the highest possible velocity to focus on muscle power. The exercises, selected to emphasize functional movements relevant to daily activities.
  Interventions: Other: Power-focused resistance training

INTERVENTIONS:
Other: Power-focused resistance training — Participants will undergo 10 weeks of power-focused resistance training.
  Other Names: Power training

SUMMARY:
Post-stroke deficits are highly common and functional impairment persists throughout life after stroke. Skeletal muscle mass and strength are fundamental contributors to mobility throughout the adult life course. Stroke-related muscle atrophy contributes to loss of strength, and declines in lower extremity function, cardiorespiratory fitness, and walking independence and post-stroke sarcopenia. Improving the quantity and function of skeletal muscle needs to be an important therapeutic target after stroke. Resistance exercise training (RET) has been shown to increase skeletal muscle mass, strength and power, reduce oxidative stress, improve cardiac function, and better regulate lipids after stroke. However, the feasibility and the effects of a power focused RET program for individuals with stroke need to be examined.

DETAILED DESCRIPTION:
This study is a single-group, open label trial examining the feasibility and preliminary effect estimates of a 10-week power-focused exercise training program in people living with stroke. Fifteen participants with chronic stroke will participate in the exercise program 3 times per week for 10 weeks at a progressive intensity. The program will take place at a community exercise gym built for older adults and people with physical disabilities. Feasibility outcomes will be assessed throughout the trial. Effectiveness outcomes will be assessed at baseline and immediately post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* ≥6 months post-stroke
* Able to walk >10 meters with or without the use of an assistive device
* Living in the community
* Mild to moderate stroke severity (modified Rankin Scale ≤3)

Exclusion Criteria:

* Any contraindications to exercise for people with cardiovascular disease, such as unstable angina, uncontrolled hypertension, orthostatic blood pressure with exercise, or uncontrolled arrhythmias
* Significant cognitive impairment that would preclude safe exercise participation (Montreal Cognitive Assessment score <26)
* Actively engaged in stroke rehabilitation services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Feasibility: Participant recruitment | Through study completion, over 13 months
  Recruitment rates (n/week) and the number of recruited subjects (n) will be reported. Criteria for success include recruitment of ≥1 participant per month and n=15 recruited in ≤13 months.
Feasibility: Sex and gender distribution | Through study completion, over 13 months
  Recruitment of males and females, men, women and gender diverse participants will be recorded (n, %). Criteria for success is <60% (n<9) of any sex or gender identity.
Feasibility: Attendance and attrition | Through study completion, over 13 months
  Percentage of sessions attended (%) and lost to follow-up (n) will be reported. Criteria for success includes ≥85% sessions attended and ≤10% (n<2) lost to follow-up.
Feasibility: Serious and non-serious adverse events | Through study completion, over 13 months
  Number of adverse events (i.e., deaths, serious and non-serious adverse events, n) will be reported. Criteria for success is 0 deaths or serious adverse events and <5 non-serious adverse events.
Feasibility: Exercise tolerance | Through study completion, over 13 months
  Adherence to the prescribed exercises (%) and abnormal blood pressure responses to exercise (n) will be recorded. Criteria for success includes ≥85 of participants performing ≥85% of sets at the prescribed intensity, and ≤25% of weeks experiencing ≥1 abnormal blood pressure response (SBP ≥210 or ≥190 for males and females, respectively).
Feasibility: Satisfaction | Immediately post-intervention (week 10)
  Satisfaction will be measured with a 5-point Likert scale (1 = not at all satisfied, 2 = not satisfied, 3 = neither satisfied or not satisfied, 4 = satisfied, and 5 = completely satisfied). Criteria for success is ≥85% of participants reporting being satisfied or completely satisfied with the program.

SECONDARY OUTCOMES:
Timed up and go test | Baseline (week 0) and post-intervention (week 10)
  The TUG is a measure of functional mobility. A standard chair (~46cm in height) will be placed at the start of a flat walking course and a cone will be placed 3 meters from the chair. Participants will stand from the chair, walk 3 meters, turn back towards the chair, and sit back down, without assistance. The task will be timed and measured in seconds.
Short physical performance battery | Baseline (week 0) and post-intervention (week 10)
  The SPPB involves 3 tests, each measuring different constructs of physical function: (1) balance (tandem stand test), (2) walking ability (4-meter walk test), and (3) lower-limb strength and endurance (5-times sit to stand test). Two trained study staff members will concurrently assess each measure. Each test on the SPPB is scored separately on a scale ranging from 0 to 4, per instrument scoring guidelines. Raw and SPPB scores will be measured.
30-second chair stand test | Baseline (week 0) and post-intervention (week 10)
  The 30sCST is a measure of lower extremity strength and endurance. A ~43cm chair with a straight back and no armrests will be placed against the wall. Participants will cross their arms and keep feet flat on the floor. With their back straight, stand up and sit down as many times as possible in 30 seconds.
Isokinetic power | Baseline (week 0) and post-intervention (week 10)
  Upper- and lower-extremity muscle power (Watts/kg) will be measured using an isokinetic dynamometer, bilaterally, at 3 different velocities (30º, 60º, 120º per second).
Isokinetic torque | Baseline (week 0) and post-intervention (week 10)
  Upper- and lower-extremity muscle torque (Nm) will be measured using an isokinetic dynamometer, bilaterally, at 3 different velocities (30º, 60º, 120º per second).
Isometric strength | Baseline (week 0) and post-intervention (week 10)
  Maximal isometric knee and elbow flexor and extensor strength (kg) and grip strength (kg) will also be measured, using a handheld dynamometer.
Global physical activity questionnaire | Baseline (week 0) and post-intervention (week 10)
  The global physical activity questionnaire (GPAQ) consists of 16 items, which are grouped to capture different domains of physical activities including work, transport and discretionary (i.e., leisure or recreational) activities. The GPAQ score may range from 0 to 80,640 MET-minutes per week, although the maximum value is likely not possible to be attained. Higher values indicate greater physical activity levels.
Stroke-Impact Scale (SIS-3.0) | Baseline (week 0) and post-intervention (week 10)
  Version 3 of the Stroke-Impact Scale (SIS-3.0) will be used to assess stroke-specific health-related quality of life. The SIS-3.0 consists of 59 items that measure 8 different domains of health: strength, hand function, (instrumental) activities of daily living, mobility, communication, emotion, cognition, and participation. Each domain is scored separately and range from 0 to 100. Higher values indicate greater health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Rehabilitation Science, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided